CLINICAL TRIAL: NCT01071187
Title: Investigation of the Efficacy and Safety of Varenicline in the Postacute Treatment of Alcohol Dependence - a Prospective, Double-blind, Placebo-controlled, Randomised Phase-II Study
Brief Title: Varenicline for Alcohol Dependence
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Pfizer (Industry)
Responsible Party: PD Dr. Christoph Fehr, Department of psychiatry and psychotherapy, university medical center of the Johannes Gutenberg-university Mainz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009-08-17; 2009-015537-67 (EudraCT Number)
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2010-09

CONDITIONS: Alcohol Dependence
Keywords: alcohol dependence; addiction; alcohol; relapse prevention
MeSH Terms: conditions — Alcoholism; Behavior, Addictive | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Experimental): Treatment with varenicline with 0,5mg daily on day 1-3, 1mg daily on day 4-7 and 2mg daily on day 8-84.
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — Varenicline 0,5mg daily on day 1-3, Varenicline 1mg daily on day 4-7 and Varenicline 2mg on day 8-84.
  Arms: Varenicline
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The varenicline for alcohol dependence trial investigates the efficacy of varenicline versus placebo for maintaining abstinence in the postacute treatment of alcohol dependent subjects. The main study hypothesis is that subjects treated with varenicline have more abstinent days during the study.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of alcohol dependence according to DSM IV
* inpatient or outpatient
* last alcohol consumption within 7-21 days before randomisation
* subjects must have gone through a detoxification program and must be free of withdrawal symptoms at randomisation
* diagnosis of nicotine dependence according to DSM IV
* sufficient knowledge of the german language
* subject is able to follow verbal and written instructions
* subject is enabled to consent
* ability of subject to understand character and individual consequences of the clinical trial
* signed and dated informed consent of the subject must bei available before start of any specific trial procedures
* subject must have a clearly stated desire to stay abstinent
* women who are postmenopausal for more than two years or women with childbearing potential who practicing two years can participate in the study

Exclusion Criteria:

* alcohol withdrawal delirium during last alcohol detoxification
* alcohol induced dementia
* severe renal insufficiency
* detoxification against subject's will
* women who are pregnant or breastfeeding or planning to become pregnant during the trial
* women with childbearing potential who not practicing a medically accepted contraception during the trial
* subjects with a known psychiatric disorder requiring treatment including a major depressive disorder, a substance dependence or abuse (besides nicotine, alcohol and cannabis)a psychosis or a dissocial personality disorder according to DSM-IV
* elevated suicide risk, defined as one positive question in the suicide section of the Mini-International Neuropsychiatric Interview (M.I.N.I.)
* subjects with acute depression, defined as a HAMD17 (german version) sum score > 9 or a BDI (german version) sum score > 12
* clinically relevant acute or chronic progressive neurologic, gastrointestinel, cardiovascular, hepatic, renal, hematological, endocrine, dermatological or respiratory disease
* severe infection, a alcohol-induced hepatitis or a uncontrolled arterial hypertension
* use of any medication that can effect on alcohol consumption within 14 days of study initiation including antidepressants, antipsychotics, anticonvulsives, benzodiazepines (besides given in the contect of the detoxification program, anticraving drugs as naltrexone, acamprosate and disulfiram and nicotine substitutes
* subjects with following lab parameters: AST upper fivehold normal limit, PTT < 50%, leucocytes <2/nl, haemoglobin < 9g/dl, thrombocytes < 80/nl, creatinine > 1,5mg/dl and creatinine clearance < 30ml/min
* history of cancer in 5 last years
* known allergy against ingredient of study drug
* history of myocardial infarction or stroke
* participation in a clinical trial during last 90 days prior to screening
* clinically relevant visual disturbance or ear disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Number of total alcohol abstinent days during he 12 weeks study period, percentage of the treatment days | 12 weeks

SECONDARY OUTCOMES:
Time in days to first alcoholic drink, assessed by the time-line-follow-back-interview | 12 weeks
Proportion of abstinent patients during the study, percentage of all patients | 12 weeks
Number of standard drinks per drinking day, assessed by the time-line-follow-back-interview. | 12 weeks
Time in days to first heavy drinking, assessed by the time-line-follow-back-interview. | 12 weeks
Number of days with heavy drinking as percentage of all treatment days, assessed by time-line-follow-back-interview. | 12 weeks
Changes in gamma-glutamyl transpeptidase levels | 12 weeks
Occurrence of adverse events | 12 weeks
Compliance of the subjects | 12 weeks
alcohol craving assessed by the obsessive compulsive drinking scale (OCDS) and a visual analog scale (VAS) | 12 weeks
Severity of the alcohol dependence assessed by the European Addiction Severity Index (EuropASI) | 12 weeks
Absolute change in the Clinical Global Impression of Change (CGI) | 12 weeks
Quality of life, assessed by the questionnaire for health condition Fragebogen zum allgemeinen Gesundheitszustand (SF-12) | 12 weeks
Number of cigarettes per day | 12 weeks
Number of nicotine abstinent days, percentage of the treatment days | 12 weeks
Severity of the nicotine dependence, assessed by the Fagerstrom test for nicotine dependence | 12 weeks
Intensity of depressive symptoms, assessed by the Beck Depression Inventors (BDI) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fehr Christoph, PD Dr., Principal Investigator — Department of psychiatry and psychotherapy, university medical center mainz of the Johannes Gutenberg-university mainz
Locations (2):
- Germany (2):
  - Department of psychiatry, psychosomatics and psychotherapie, Markus hospital, Frankfurt am Main, Frankfurt am Main, Hesse
  - Department of psychiatry and psychotherapy, University medical center of the Johannes Gutenberg.university Mainz, Mainz, Rhineland-Palatinate